CLINICAL TRIAL: NCT06885125
Title: Randomized Controlled Study on the Effect of a DietAry interveNtion in Ameliorating fertiliTy Parameters in Women With endomEtriosis Undergoing IVF (The DANTE Study)
Brief Title: Dietary Intervention to Improve Fertility in Women With Endometriosis Undergoing IVF
Acronym: DANTE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: UNIVERSITE CATHOLIQUE DE LOUVAIN (Unknown); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); University of Edinburgh (Other); STICHTING RADBOUD UNIVERSITAIR MEDISCH CENTRUM (Unknown); UNIWERSYTET MEDYCZNY W LUBLINIE (Unknown); SVEUCILISTE U ZAGREBU MEDICINSKI FAKULTET (Unknown); University College Cork (Other); Endometriosis UK (Unknown); Wageningen University (Other); Endometriose Stichting (Unknown); Belgian Volition SRL (Unknown); ASSOCIATION OF PEOPLE WITH ENDOMETRIOSIS I AM 1 IN 10 (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DANTE Study
Record Dates: First submitted 2025-02-05; First posted 2025-03-20 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-01

CONDITIONS: Endometriosis
Keywords: IVF; endometriosis; anti-inflammatory diet
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The treatment will be kept blind for both the medical and laboratory personnel performing the in vitro fertilization procedures. The allocation branch will be revealed to the data manager at the end of data collection related to the primary outcome.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-Inflammatory Diet (Experimental): Patients will follow a 12-week anti-inflammatory diet, followed by the standard IVF treatment protocol.
  Interventions: Dietary Supplement: anti-inflammatory diet
- Controls (No Intervention): Patients will undergo the standard IVF treatment protocol without any dietary intervention.

INTERVENTIONS:
Dietary Supplement: anti-inflammatory diet — The anti-inflammatory diet consists of a 12-week plant-based diet, followed by guidance and monitoring from a nutritionist.
  Arms: Anti-Inflammatory Diet

SUMMARY:
The goal of this randomized controlled trial is to assess whether a 12-week anti-inflammatory diet can improve fertility outcomes in women with endometriosis undergoing In Vitro Fertilization (IVF).

The main questions are:

* Does the anti-inflammatory diet reduce the rate of inadequate ovarian response to hormonal stimulation (retrieval of ≤3 oocytes)?
* Does it improve secondary outcomes such as embryo quality, pregnancy rates, inflammation markers, and quality of life?

Researchers will compare two groups:

* Women receiving standard IVF protocols.
* Women undergoing the same IVF protocol plus the anti-inflammatory diet.

Participants will:

* Be randomized into one of the two groups.
* Follow dietary counseling sessions and complete dietary assessments (diet group).
* Provide biological samples (e.g., plasma, vaginal and fecal swabs, and follicular fluid) before and after the dietary intervention to evaluate potential differences in inflammation, hormonal levels, and microbiome composition between the two groups and across timepoints (pre- and post-diet).
* Complete questionnaires on quality of life, sexual function, and symptomatology severity before and after the intervention to assess differences between the two groups and across timepoints.

DETAILED DESCRIPTION:
Women who agree to participate in the study will be randomized into two groups: one group will receive standard IVF protocols, and the other will undergo a 12-week anti-inflammatory diet followed by the standard IVF protocol. In both groups, participants' dietary habits will be monitored throughout the study period to detect any variations. The primary outcome will be to compare the rate of inadequate ovarian response to hormonal stimulation (defined as the retrieval of ≤3 oocytes according to the Poseidon 2016 criteria) in infertile women with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Age < 40 years
* Pregnancy seeking for more than 12 months
* Regular menstrual cycle, i.e. mean cycle interval between 21 and 35 days
* Ultrasonographic diagnosis of ovarian endometriomas or deep peritoneal endometriosis.
* Antral Follicle Counts (AFC) ≥ 5 (no other cause of reduced ovarian reserve).
* Absence of ureteral stenosis or intestinal subocclusive symptoms

Exclusion Criteria:

* Contraindication to pregnancy
* Hydrosalpinx
* Endometriomas with a mean diameter > 4 cm
* Submucosal fibroids or large intramural or subserosal fibroids (≥ 5 cm).
* Doubtful sonographic findings that do not allow to reliably rule out malignancy.
* severe male factor (<1 million sperm/ml)

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 438 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Inadequate ovarian response | During the oocyte retrieval procedure
  Rate of inadequate ovarian response to hormonal stimulation (defined as the retrieval of ≤3 oocytes according to the Poseidon 2016 criteria) in infertile women with endometriosis who follow an anti-inflammatory diet compared to those who do not follow any specific diet.

SECONDARY OUTCOMES:
Adherence to the intervention | 3 months
  Adherence to the intervention using 24 hour recall.
Fertilisation rate | The day after oocyte retrieval
  Fertilisation rate per aspirated oocyte retrieved. Defined as the appearance of 2 pronuclei (PN)
Embryo quality | Up to six days after oocyte pick-up
  Good quality blastocysts according to Gardner classification
Cumulative pregnancy rates | 12 months
  All clinical pregnancies achieved by IVF, including the transfer of fresh embryos and all cryopreserved-thawed embryos from the stimulation cycle.
Miscarriage rate | 24 months
  Spontaneous or planned abortions.
Cumulative Live Birth Rate | 24 months
  All live birth achieved by IVF, including the transfer of fresh embryos and all cryopreserved-thawed embryos from the stimulation cycle.
Microbiome composition | 4 months
  The difference in microorganism species distribution according to 16S RNA sequencing analysis between the control group and the study group, as well as before and after the diet in the study group. Both the vaginal and gut microbiome will be analyzed.
Concentration of Steroid Hormones | 4 months
  The difference between the steroid cascade in follicular fluids of women following the diet and those not following the diet, specifically focusing on the following hormones: Aldosterone, Cortisol, Cortisone, 11-DeoxyCortisol, 21-DeoxyCortisol, Corticosterone, 11-Deoxycorticosterone, DHEAS, DHEA, Estradiol, Androstenedione, Testosterone, DHT, 17-OHProgesterone, and Progesterone.
Inflammation Index | 4 months
  The difference in the inflammation index between the control group and the study group, as well as pre- and post-diet changes within the study group, will be evaluated using a composite blood-based inflammation index called the INFLA-score. This index is based on four circulating biomarkers-C-reactive protein (CRP) levels, blood platelet count (Plt), white blood cell count (WBC), and granulocyte-to-lymphocyte ratio (GLR)-and captures both serum and cellular-circulating inflammation.
Quality of life (using 30-item Endometriosis Health Profile) | 4 months
  Quality of life differences between the control group and the study group, as well as pre- and post-diet changes within the study group, will be evaluated using the Endometriosis Health Profile-30 (EHP-30) questionnaire. The EHP-30 consists of 30 items divided into five subscales: 'pain,' 'control and powerlessness,' 'social support,' 'emotional well-being,' and 'self-image.' Each subscale is standardized on a scale from 0 to 100, where lower scores indicate better quality of life.
Sexual function (using Female Sexual Function Index) | 4 months
  Sexual function differences between the control group and the study group, as well as pre- and post-diet changes within the study group, will be evaluated using the Female Sexual Function Index (FSFI), a questionnaire with a score range from 2 to 36, where higher scores indicate better sexual function.
Symptomatology severity (using Numeric Rating Scale) | 4 months
  Symptomatology severity differences between the control group and the study group, as well as pre- and post-diet changes within the study group, will be evaluated using Numeric Rating Scale (NRS, min 0-max 10), where higher scores indicate worse symptom severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vigano P, Abodi M, Benaglia L, Bolis I, Casalechi M, Ferraro C, Li Piani L, Reschini M, Ruggiero F, Salmeri N, Somigliana E, Horne AW, Nap AW, Dolmans MM; EUmetriosis Working Group. Effectiveness of an anti-inflammatory diet before in vitro fertilisation in women with endometriosis: protocol for a randomised controlled trial. BMJ Open. 2025 Dec 23;15(12):e108596. doi: 10.1136/bmjopen-2025-108596. PMID 41436256